CLINICAL TRIAL: NCT06298851
Title: Comparative Effects of Lower Body Quadrant Neural Mobilization and Stretching in Collegiate Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-772.02-2026
Record Dates: First submitted 2024-02-23; First posted 2024-03-07 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Sports Physical Therapy; Stretch; Stretch Injury
Keywords: football players; neural mobilization; static stretching; dynamic stretching

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neural Mobilization Group (NMG) (Experimental): Participants of NMG performed sciatic, femoral and peroneal nerve and lumbar region gliding. All glides include 4 sets of 10 repetitions, with each gliding cycle lasting 6 seconds, and a 1-minute rest between sets for both extremities.
  Interventions: Other: Neural Mobilization Group (NMG)
- Dynamic Stretching Group (DSG) (Experimental): 4 sets of 10 repetitions will be performed, each exercise cycle lasting 6 seconds, and a 1-minute rest period will be given between sets. All stretching exercises will be performed in two circuits.
  Interventions: Other: Dynamic Stretching Group (DSG)
- Static Stretching Group (SSG) (Experimental): 4 sets of 4 repetitions will be applied to the lumbar extensor, hamstring, quadriceps and gastrocnemius muscles located in both extremities, each stretching will last for 15 seconds and a 1-minute rest period will be given between sets.
  Interventions: Other: Static Stretching Group (SSG)

INTERVENTIONS:
Other: Neural Mobilization Group (NMG) — Femoral nerve gliding: Mobilization of the femoral nerve will performed while the participant in the prone position and the hip hyperextended. Tension will applied by placing the knee in full flexion and the ankle in plantar flexion.
  Sciatic nerve gliding: Participants will take turns while sitting with the trunk in thoracic flexion; perform knee extension/dorsiflexion with cervical extension and knee flexion/plantar flexion with cervical flexion. Tension will applied by flexing the hip and dorsiflexing the ankle to the point where stress will felt.
  Peroneal nerve gliding: The participant will asked to maintain this position in a supine position by placing the ankle in inversion and plantar flexion. From a starting position consisting of ankle dorsiflexion, knee, and hip extension, the patient will return to the starting position by simultaneously performing ankle plantar flexion and inversion, full knee flexion, and 90 degrees of hip flexion.
  Arms: Neural Mobilization Group (NMG)
Other: Dynamic Stretching Group (DSG) — Exercises will include functional activities that provided dynamic stretching of the hamstrings, quadriceps, hip flexor, extensor, abductor and adductor muscles, and gastrosoleus muscle. All stretching exercises will be performed in two circuits in an area of 15 m2. 4 sets of 10 repetitions will be performed, each exercise cycle lasting 6 seconds, and a 1-minute rest period will be given between sets. This process will be repeated for both extremities.
  Arms: Dynamic Stretching Group (DSG)
Other: Static Stretching Group (SSG) — Static stretching exercises will be described to the participants as given below:
  Standing quadriceps stretch: The participant will stand upright, fold one knee and bring the heel towards the buttock while holding the foot with one hand.
  Modified hamstring stretching: The participant will be in a seated position with one leg straight and will place the other foot on the inside of the straight leg and reach forward.
  Gastrocnemius stretching: The participant stands with feet 60-90 cm from the wall, leaning against the wall with both hands, keeping the back leg straight and the front leg slightly bent.
  Adductor stretching: Participants will be in a sitting position with an erect spine, bending and releasing their knees with the soles of their feet touching.
  Lumbar stretching: In a sitting position, participants keep one leg straight and place the other foot on the outside of the straight leg and rotate the body diagonally.
  Arms: Static Stretching Group (SSG)

SUMMARY:
Neural mobilization (NM) refers to a therapeutic interventions that aim to directly or indirectly influence neural structures and adjacent tissues through manual techniques or exercise. The application of NM has been investigated in both patients and healthy individuals. In this study, participants from an amateur football team will be allocated into three groups, each undergoing pre-training warm-up protocols incorporating NM, dynamic stretching, or static stretching. Following the warm-up protocols, the effects on flexibility and athletic performance will be evaluated and compared across the groups.

DETAILED DESCRIPTION:
Neural mobilization (NM) is an intervention that involves manual techniques or exercises designed to affect neural structures and surrounding tissues. It aims to restore normal neural mechanical and physiological responses to movement and posture by facilitating the sliding and tension of the nerves. NM techniques can be divided into two groups: gliding, which involves different joint movements, and tension, which extends the nerves in more than one joint. Although NM has been linked to various neurophysiological benefits, the precise mechanisms underlying its clinical efficacy remain uncertain.

The peripheral nervous system demonstrates the ability to adapt to changing mechanical forces encountered during daily activities and sports through nerve gliding and sliding mechanisms. Impaired gliding may result in increased neural stress and ischemic damage, affecting neural function. NM has been shown to improve lower extremity flexibility, which is crucial for enhancing functionality and minimizing injury risk in athletes. Neurodynamic techniques are frequently used to increase hamstring flexibility and reduce neural mechanosensitivity, contributing positively to athletic performance and injury prevention.

The aim of this study is to examine the comparative effects of static stretching, dynamic stretching and neural mobilization techniques used in pre-training warm-up sessions on flexibility and performance in collegiate football players.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25
* Not having had a lower or upper extremity injury in the last 3 months
* Not having had surgery in the last 6 months
* Playing amateur football regularly for at least 1 year

Exclusion Criteria:

* Orthopedic, neurological, rheumatological or cardiorespiratory health problems that would prevent them from performing the tests

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Straight Leg Raise Test | From pre-interventional time to post-interventional about an hour
  The passive straight leg raise test will be used to determine changes in the flexibility of the hamstring muscle. With the participant in the supine position, the lateral condyle of the femur, fibular head, and fibular malleolus will be identified. The axis of a goniometer will be placed over the protrusion of the greater trochanter of the femur. One of the arms of the goniometer will be placed parallel to the table. The knee and ankle will be kept in the extension position. By holding the talus and without rotating the hip, flexion of the hip will be gradually increased. Participants' lower extremities will be elevated until they complain of pain in the rear thigh area. Care will be taken to ensure that they do not bend their knees and that the pelvis is not in retroversion. Then, the other arm of the goniometer will be placed in the direction of the line between the head of the fibula and the fibular malleolus and the degree of height of the straight leg will be noted.

SECONDARY OUTCOMES:
Y Balance Test | From pre-interventional time to post-interventional about an hour
  Participants will stand on the foot plate in the center of the Y Balance Test area. Participants will be instructed to maintain a single-leg stance while reaching as far as possible with the opposite leg and return to the starting position on the middle platform without losing balance. In the test, participants will be allowed 3 attempts for both lower extremities and will be asked to reach the maximum distance in 3 directions anterior, posteromedial and posterolateral. The maximum reach distance will be recorded for each consecutive attempt.

OTHER OUTCOMES:
One-Leg Forward Jump Test | From pre-interventional time to post-interventional about an hour
  A 2-meter tape measure will be placed on a flat surface for the test. Participants will be asked to stand on one leg with their toes remaining at zero on the tape measure, jump forward as much as possible with their hands on their waist, and land on the same foot. The place where he places his fingertip after jumping will be recorded by reading from the tape measure. Participants will be informed that they must maintain their position for 2 seconds after landing. The test will be applied separately for dominant and non-dominant feet. Participants will be given 1 trial application, followed by 3 tests and the best result will be recorded in centimeters. There will be a 30-second rest between tests.
T Test | From pre-interventional time to post-interventional about an hour
  The T test consists of 4 contact points formed in a T shape in an area of 10 meters long and 10 meters wide. In this test, the aim is to complete a series in the shortest time that requires the participant to move in different directions and in different ways between these contact points, and the participant always looks in the same direction. The participant will change direction by stepping forward, backward, right and left. This test requires covering a total distance of 40 meters, including 10 m forward, 10 m to the right, 10 m to the left and 10 m back.
BlazePod Reaction Time Determination Test | From pre-interventional time to post-interventional about an hour
  The BlazePod test, utilizing sensor-equipped pods will assess reaction time by measuring reflexes and instantaneous speed. For lower extremity evaluation, three pods will be mounted on a wall 1.5 m above the floor and 1.5 m apart. Positioned 3 meters away from the wall, athletes will respond to random light signals by running and touching the illuminated compartment. Each trial will consist of 6 light triggers, with 2 trials performed and a 3-minute rest between trials. Performance will be evaluated based on the number of touches, reaction time, and average reaction time over 15 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)